CLINICAL TRIAL: NCT03386552
Title: A Randomized, Double Blind, Controlled, Parallel Groups, Multi-center Phase II Clinical Study of Lidocaine Pertubation as a Treatment for Couples With Unexplained Infertility
Brief Title: A Study of Lidocaine Pertubation as a Treatment for Unexplained Infertility
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isifer AB (Industry)
Collaborators: Ferring Pharmaceuticals (Industry); Vinnova (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISI-2015-1
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Buffers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isifera+ (Experimental): Subjects are pertubated with Isifer+ solution containing lidocaine 0.5 mg/ml
  Interventions: Drug: Isifera+
- Buffer (Placebo Comparator): Subjects are pertubated with a buffer solution without lidocaine
  Interventions: Drug: Buffer

INTERVENTIONS:
Drug: Isifera+ — Pertubation solution of lidocaine 0.5 mg ml in Ringer-Acetate buffer
  Arms: Isifera+
Drug: Buffer — Pertubation solution of Ringer-Acetate buffer
  Arms: Buffer

SUMMARY:
The present investigation is evaluating a method for improving pregnancy outcome of couples with unexplained infertility. The method utilizes an adjuvant pre-treatment prior to insemination, that is pertubation, i.e. flushing the uterus and fallopian tubes before insemination with a specially developed solution with the aim to increase fertility. The clinical trial is a phase II double blind, randomized, controlled and multi-center trial .

DETAILED DESCRIPTION:
Couples interested in participating in the clinical study must have undergone a complete investigation for their infertility and have at least one year of unsuccessful attempts to achieve pregnancy. Following inclusion in the study, patients will be monitored with vaginal ultrasound to ensure a leading follicle of at least 18 mm.The subjects with one or two follicles ≥18 mm will be given Ovitrelle® (Merck), dose 250 ug (6500 IU) of Human Chorionic Gonadotropin (HCG), subcutaneously for ovulation induction. 12-24 h after the HCG injection, patients will be randomized and pertubated with either test or control solution.

12 -24 hours after the pertubation insemination (IUI) will be given to all patients. A blood sample is taken 14-17 days after IUI, for analysis of serum HCG level and possible pregnancy. In case of positive answer a second confirmatory sample will be obtained 48-72 hours later. In case of confirmed elevated HCG, the clinical pregnancy (CP) will be assessed with vaginal ultrasound examination 6-7 week after IUI. Baby take home rate data will be collected for couples with clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Females with, unexplained infertility, 20-38 years of age. Normal menstrual cycle length of 26-35 days, male partner 20-70 years of age, Duration of infertility should have lasted more than one year and subject should have signed informed consent.

Couples must fulfil all laboratory tests for inclusion, negative HIV-1, HCV, HBV, CMV virology, chlamydia and syphilis. For female also negative toxoplasmosis, rubella and hormonal screen within normal range. Furthermore patent fallopian tubes should be confirmed by ultrasound hysterosalpingography and males should present a normal semen analysis

Exclusion Criteria:

Continuous treatment with NSAID, corticosteroids or other drugs, which can cause an increased risk of infection, clinical signs of PID, known hypersensitivity to local anaesthetics, non-patent fallopian tubes, abnormal uterine cavity, submucous myoma > 2 cm in diameter, any disease or laboratory finding considered of importance by the investigator not to include the patient, laparoscopically confirmed endometriosis of greater severity than mild, endometriosis of any severity with adhesions. More than 2 previous inseminations or previous unsuccessful IVF treatment.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | day 14-17 after IUI
  serum-HCG

SECONDARY OUTCOMES:
Baby take home rate | At delivery / Miscarriage
  Delivery of baby

CONTACTS AND LOCATIONS:
Overall Officials: Jack Spira, Md PhD, Study Chair — Isifer AB
Locations (1):
- InviMed-T sp. z o.o, Warsaw, Poland

REFERENCES:
- [Result] Edelstam G, Sjosten A, Bjuresten K, Ek I, Wanggren K, Spira J. A new rapid and effective method for treatment of unexplained infertility. Hum Reprod. 2008 Apr;23(4):852-6. doi: 10.1093/humrep/den003. Epub 2008 Feb 15. PMID 18281242
- See also: A new rapid and effective method for treatment of unexplained infertility. — https://www.ncbi.nlm.nih.gov/pubmed/18281242